CLINICAL TRIAL: NCT01153607
Title: Open-label, Non-randomized, Multicenter Positron Emission Tomography (PET) Imaging Study to Evaluate a Single Dose of BAY1006578 for Its Diagnostic Potential in Discriminating Patients With Probable Alzheimers Disease From Healthy Volunteers and to Evaluate the Radiation Dosimetry of a Single Dose of BAY1006578 in Healthy Volunteers
Brief Title: Evaluation of the Diagnostic Potential of BAY1006578 in Probable Alzheimers Disease Patients Versus Healthy Volunteers and Radiation Dosimetry of BAY1006578 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Life Molecular Imaging SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14708; 2009-017166-24 (EudraCT Number)
Record Dates: First submitted 2010-04-23; First posted 2010-06-30 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Diagnostic Imaging
Keywords: Alzheimer's disease; Diagnostic imaging; PET diagnosis; PET tracer
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: BAY1006578
- Arm 2 (Experimental)
  Interventions: Drug: BAY1006578
- Arm 3 (Experimental)
  Interventions: Drug: BAY1006578

INTERVENTIONS:
Drug: BAY1006578 — Alzheimer Disease patients: Single intravenous bolus injection of 250 MBq BAY1006578 on day one of the treatment period, PET
  Arms: Arm 1
Drug: BAY1006578 — Healthy volunteers for brain imaging: Single intravenous bolus injection of 250 MBq BAY1006578 on day one of the treatment period, PET
  Arms: Arm 2
Drug: BAY1006578 — Healthy volunteers for whole body imaging: Single intravenous bolus injection of 190 MBq BAY1006578, whole body PET for evaluation of effective dose, kinetics of BAY1006578 in blood
  Arms: Arm 3

SUMMARY:
PET (positron emission tomography) imaging with BAY1006578 for investigation of diagnostic potential in probable Alzheimer Disease patients versus healthy volunteers and radiation dosimetry in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* All:

  * Males or females aged >/- 50 years
  * Participants must be able to understand the information provided on purpose and conduct of the clinical study, must be capable of giving fully informed consent in writing, and have read and signed the informed consent prior to study participation
* Healthy volunteers for brain imaging:

  * Mini-Mental State Examination (MMSE) score of >/= 28
  * CDR score of zero (0)
* Patients for brain imaging:

  * Patient fulfills Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) and National Institute of Neurological and Communicative Disorders and Stroke, Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria for probable Alzheimer's Disease (AD), which are cognitive deficits such as memory decline and impairment in at least one other cognitive domain (e.g. aphasia, apraxia, agnosia or executive dysfunction)
  * Patient has mild to moderate dementia with a dementia score of >/= 20 on the Mini Mental State Examination (MMSE) / with a Clinical Dementia Rating score of 1 or 2 (CDR)

Exclusion Criteria:

* All:

  * No significant disease or drug use
* Patients for brain imaging:

  * Evidence for any other neurological or psychiatric disease
* Healthy volunteers for brain imaging:

  * Family history of Alzheimer's Disease in a 1st or 2nd degree relative under 75 years of age

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Discrimination of probable Alzheimer's Disease patients from healthy volunteers by BAY1006578 brain Positron Emission Tomography (PET) imaging as evaluated by different quantification approaches | Day 1 - day of study tracer administration

SECONDARY OUTCOMES:
Discrimination of probable Alzheimer's Disease patients from healthy volunteers by BAY1006578 brain Positron Emission Tomography (PET) imaging as evaluated by visual analysis and by standard parameters (e.g. Standardized Uptake Values=SUV) | Day 1 - day of study tracer administration
Electrocardiogram (ECG) | At least once within 8 days after treatment
Blood pressure | At least 2 times within 8 days after treatment
Adverse events collection | Continuously and for a maximum of 28 days after end of observation phase

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Turku, Finland
- Stockholm, Sweden